CLINICAL TRIAL: NCT06517277
Title: Retrospective Hospital Study of Haemophilus Influenzae Pneumonia in Adults: Relapse and Severity
Brief Title: Haemophilus Influenzae Pneumonia in Adults
Acronym: REHALIgraviTY
Status: Completed | Type: Observational
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Collaborators: URC-CIC Paris Descartes Necker Cochin (Other)
Responsible Party: Sponsor
Other Study IDs: APHP240446
Record Dates: First submitted 2024-07-18; First posted 2024-07-24 (Actual); Last update posted 2025-09-12 (Actual); Status verified 2025-09

CONDITIONS: Haemophilus Influenzae Pneumonia
Keywords: Haemophilus influenzae pneumonia; Adult patients; Relapse of Haemophilus influenzae pneumonia; Severity of Haemophilus influenzae pneumonia; Antibiotic resistance profiles of Haemophilus influenzae strains; Chest radiological patterns

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Patients: Hospitalized patients for a Haemophilus influenzae pneumonia in 13 AP-HP hospitals between 09/01/2022 to 08/31/2023.
  Interventions: Other: Collection of data from the patient's medical file

INTERVENTIONS:
Other: Collection of data from the patient's medical file — Collection of data from the patient's medical file. Relapses will be collected up to 3 months after Haemophilus influenzae pneumonia first episode.

SUMMARY:
Haemophilus influenzae is a Gram-negative coccobacillus capable of colonizing and infecting the human respiratory tract.

In the adult population, patients with an abnormality of their mucociliary epithelium and a deficiency in innate or adaptive immunity are particularly exposed.

The Infectious and Tropical Diseases department of Necker-Enfants Malades hospital has noted a recent increase in the number of cases of respiratory infections due to H. influenzae, with a high frequency of early relapses and recurrences despite appropriate treatment.

The research focuses on lower respiratory infections (pneumonia) caused by Haemophilus influenzae in adults, excluding pneumonia acquired under mechanical ventilation linked to Haemophilus influenzae in patients in 13 AP-HP hospitals during 12 months, from 09/01/2022 to 08/31/2023.

DETAILED DESCRIPTION:
Haemophilus influenzae is a Gram-negative coccobacillus capable of colonizing and infecting the human respiratory tract.

In the adult population, patients with an abnormality of their mucociliary epithelium and a deficiency in innate or adaptive immunity are particularly exposed.

The Infectious and Tropical Diseases department of Necker-Enfants Malades hospital has noted a recent increase in the number of cases of respiratory infections due to H. influenzae, with a high frequency of early relapses and recurrences despite appropriate treatment.

The research focuses on lower respiratory infections (pneumonia) caused by Haemophilus influenzae in adults, excluding pneumonia acquired under mechanical ventilation linked to Haemophilus influenzae in patients in 13 AP-HP hospitals during 12 months, from 09/01/2022 to 08/31/2023.

The main objective of the study is to identify factors associated with relapse in hospitalized adult Haemophilus influenzae pneumonia.

ELIGIBILITY:
Inclusion Criteria:

* Acute respiratory symptoms: cough and/or dyspnea and/or purulent sputum or worsening of the color of the sputum for patients with chronic respiratory pathology, chest pain, desaturation defined by saturation < 95% in ambient air
* Inflammatory syndrome: fever ≥ 38.5°C or CRP ≥ 30 mg/L
* Pulmonary imaging (x-ray or CT scan) compatible with pneumonia
* Good quality respiratory sample (for cytobacteriological examination of sputum (CBES) : leukocytes > 25/mm3 and cells < 10/mm3) positive in culture for H. influenzae at a significant threshold (for CBES ≥ 107 CFU/mL, for "standard" bronchial aspirate ≥ 105 CFU/mL, for protected bronchial aspiration ≥ 103 CFU/mL, for bronchoalveolar lavage ≥ 104 CFU/mL)
* Respiratory antibiotic therapy started by the clinician

Exclusion Criteria:

* Age < 18 years
* Opposition formulated (following receipt of the study information note)
* Legal protection measure (impossibility of collecting non-opposition)
* Ventilator-associated pneumonia (VAP)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Hospitalized patients for a Haemophilus influenzae pneumonia in 14 hospitals of Assistance Publique - Hôpitaux de Paris, between 09/01/2022 to 08/31/2023.
Sampling Method: Non-Probability Sample
Enrollment: 203 (Actual)
Dates: Start 2024-07-26 (Actual); Primary Completion 2024-09-01 (Actual); Study Completion 2024-09-01 (Actual)

PRIMARY OUTCOMES:
Relapse associated factors of Haemophilus influenzae pneumonia | 15 months
  Relapse associated factors with the Haemophilus influenzae pneumonia in hospitalized adult.
  Relapse of Haemophilus influenzae pneumonia defined as:
  * Definite relapse: acute respiratory symptoms (cough and/or dyspnea and/or purulent sputum), inflammatory syndrome (clinical: fever ≥ 38.5°C or biological: CRP ≥ 30 mg/L), respiratory antibiotic therapy started by the clinician, new good quality respiratory sample positive in culture for Haemophilus influenzae within 90 days following the first episode.
  * Probable relapse: acute respiratory symptoms, inflammatory syndrome (clinical: fever ≥ 38.5°C or biological: CRP ≥ 30 mg/L), respiratory antibiotic therapy started by the clinician, absence of microbiological documentation of the new episode, within 30 days following the first episode.

SECONDARY OUTCOMES:
Severity associated factors in Haemophilus influenzae pneumonia | 15 months
  Identify the factors associated with severity in Haemophilus influenzae pneumonia. Severity is defined as: oxygen therapy > 3 L/minute or need for hospitalization in intensive care unit or death.
Antibiotic resistance profiles of Haemophilus influenza strains | 15 months
  Specify the antibiotic resistance profiles of the strains of Haemophilus influenzae responsible for pneumonia during the study period.
Pulmonary radiological patterns in Haemophilus influenzae pneumonia | 15 months
  Describe the pulmonary radiological patterns associated with Haemophilus influenzae pneumonia.

CONTACTS AND LOCATIONS:
Overall Officials: Olivier LORTHOLARY, MD, PhD, Study Director — Assistance Publique - Hôpitaux de Paris
Locations (12):
- France (12):
  - Hôpital Béclère, Clamart
  - Hôpital Beaujon, Clichy
  - Hôpital Raymond Poincaré, Garches
  - Hôpital du Kremlin-Bicêtre, Le Kremlin-Bicêtre
  - Hôpital Lariboisière, Paris
  - Hôpital Saint-Louis, Paris
  - Hôpital Saint-Antoine, Paris
  - Hôpital La Pitié Salpêtrière, Paris
  - Hôpital Cochin, Paris
  - Hôpital Européen Georges Pompidou, Paris
  - Hôpital Necker-Enfants Malades, Paris
  - Hôpital Bichat, Paris

IPD SHARING:
Plan to Share IPD: No